CLINICAL TRIAL: NCT03906383
Title: Changes in the Diameter of Retinal Vessels After Remote Ischemic Conditioning in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RIK_RVA Diabetes
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Retinal Ischemia; Diabetes Complications; Ischemia; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Complications; Ischemia; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Ischemic Conditioning (Experimental)
  Interventions: Other: Remote Ischemic Conditioning

INTERVENTIONS:
Other: Remote Ischemic Conditioning — Brief reversible restriction of blood flow to upper limb in four cycles of 5 minutes of inflation at 200mm Hg followed by 5 minutes of deflation.

SUMMARY:
Remote ischemic conditioning (RIC) is a therapeutic strategy for protecting organs or tissue against the detrimental effects of acute ischemia-reperfusion injury. It remains unknown whether this can be used in retinal ischemic diseases. The purpose of the present study is to examine if the autoregulation of retinal vessel diameters in diabetic patients change after remote ischemic conditioning and if the observations are different from what have been observed in normal persons.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1
* Diabetic retinopathy

Exclusion Criteria:

* Previous treatment for diabetic retinopathy
* Other ocular and systemic diseases requiring treatment
* Pregnancy or lactation

Ages: 20 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Diameter change of retinal vessels | Immediately after and one hour after
  Diameter change from baseline in percent.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aarhus, Aarhus C, Danmark, Denmark

REFERENCES:
- [Derived] El Dabagh Y, Petersen L, Pedersen M, Bek T. Reduced baseline diameter and contraction of peripheral retinal arterioles immediately after remote ischemia in diabetic patients. Graefes Arch Clin Exp Ophthalmol. 2019 Oct;257(10):2095-2101. doi: 10.1007/s00417-019-04407-x. Epub 2019 Jul 4. PMID 31273510